CLINICAL TRIAL: NCT06629155
Title: Disentangling Cognitive Functioning and Visual Scanning Deficits in Cognitive Test Results in Multiple Sclerosis (MS)
Brief Title: Studying Eye Movement Deficits and Cognitive Impairment in Patients with Multiple Sclerosis Using Infrared Eye Tracking and Cognitive Tests
Acronym: VisuMS
Status: Not yet recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Jeroen Van Schependom, Research Professor, Universitair Ziekenhuis Brussel
Other Study IDs: 24162_VisuMS
Record Dates: First submitted 2024-10-01; First posted 2024-10-08 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis; Internuclear Ophthalmoplegia
Keywords: Cognitive impairment; Multiple Sclerosis; Internuclear Ophthalmoplegia; SDMT
MeSH Terms: conditions — Multiple Sclerosis; Ocular Motility Disorders; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- People with multiple sclerosis: This study will include 50 people with MS (see in/exclusion criteria under "Eligibility").
  Interventions: Diagnostic Test: Infrared oculography

INTERVENTIONS:
Diagnostic Test: Infrared oculography — Eye movements will be captured through infrared oculography and processed via in-house algorithms.

SUMMARY:
The goal of this observational study is to study the relationship between cognitive problems and problems in eye movements in Multiple Sclerosis (MS).

The main questions it aims to answer are:

* What is the correlation between eye movement parameters (VDI AUC and VDI Pv/Am, left and right) and SDMT scores in patients with MS?
* What is the number of patients with VDI AUC>1.174 and/or VDI Pv/Am>1.180 assessed by infrared oculography during prosaccades at 15 degrees left or right?
* What is the correlation between eye movement parameters (VDI AUC and VDI Pv/Am, left and right) and cognitive test scores in patients with MS?

Participants will perform specific cognitive tests and eye movements will be measured through infrared oculography.

The primary hypothesis for the study is: participants who exceed the treshold (VDI AUC>1.174 and/or VDI Pv/Am>1.180, left or right) will perform worse on cognitive tests compared to those who don't.

DETAILED DESCRIPTION:
As previously described in the brief summary, this clinical study aims to investigate the relationship between cognitive impairment and eye movement parameters in Multiple Sclerosis (MS).

Cognitive tests

Cognitive impairment is a common symptom in patients with MS. The most affected cognitive domains are information processing speed and visual memory, but also the domains of attention, executive function, working memory, visuospatial processing and verbal memory can be affected. There are different valid screening and evaluation tools for cognitive impairment (CI) described and used in the MS field. This clinical study will use the tests of the Brief International Cognitive Assessment for MS (BICAMS).

Infrared oculography

Another common symptom in MS is problems with eye movements. An eye condition commonly seen in these patients is internuclear ophthalmoplegia (INO). It is a specific conjugate horizontal gaze disorder characterized by slowed movement of the adducting eye relative to the abducting eye in horizontal saccades, resulting from damage to the medial longitudinal fasciculus (MLF). This may lead to (transient) diplopia or 'blurring of vision', particularly during horizontal gaze. INO can be diagnosed by using infrared oculography, a noninvasive method of quantifying eye movements. Recent research indicates that eye movements can reflect certain aspects of brain function and provide insights into cognitive impairments. Therefore, this study aims to investigate the prevalence of INO in MS using infrared oculography, compare the diagnosis of INO using infrared oculography with clinical examination by a physician and lastly explore the relationship between the presence of INO and cognitive decline.

Investigational plan

The study will be a prospective observational multi-center, cross-sectional cohort study.

Patients will be recruited at the National MS Center Melsbroek (NMSC) in close collaboration with Prof. Miguel D'haeseleer (Neurology), Prof. Daphne Kos (Rehabilitation and research coordinator) and Mieke D'hooge (Neuropsychologist). At any moment in time about 80 MS patients are in a short rehabilitation admission at the National MS Centre Melsbroek. Additionally, patients will be recruited from the MS department in the neurology wing of UZ Brussels. The MS team at UZ Brussel comprises Prof. Dr. Ir. Guy Nagels (Head of Departement), Prof. Dr. Miguel D'Haeseleer, Prof. Dr. Marie D'Hooghe, Dr. Stéphanie Hostenbach, and Annick Van Merhaegen.

When patients fulfill the inclusion criteria and give active informed consent, they will be contacted by phone to schedule their visit. If patients would like more information they can contact the investigator by phone.

During their visit, patients will undergo cognitive testing and infrared oculography. The investigators will start with the cognitive assessments, which include the BICAMS and the PASAT. The BICAMS is a 15-minute-long neuropsychological evaluation battery (9). The PASAT typically lasts 15-20 minutes. Altogether, the cognitive testing will take around 40 minutes. Following this, the infrared oculography measurements will be done. According to a study that provided a standardized and reproducible protocol for infrared oculography measurements, the total experiment duration was 21 minutes, excluding instructions. Thus, the oculography process will take roughly 30 minutes. To ensure enough time for each patient and avoid rushing, the total duration of the visit will be approximately 1,5 hours per patient.

After their first visit, there is no need for a follow-up. Should any questions arise afterward, they are welcome to reach out to us via phone or email.

Patients may withdraw from the study at any time for any reason.

Quality assurance plan/ data checks

After measurement, the variables that are needed for analysis have to be imported into Matlab. The analysis will be automated and checked for quality issues by researchers. To pass quality control, at least 50% of prosaccades at 15 degrees must be captured.

Source data verification To ensure accuracy and completeness, two researchers will evaluate and verify the source data. Any discrepancies will be documented and managed in line with the Good Clinical Practice guidelines.

Data dictionary

INO will be quantified through eye movement parameters Cognitive scores will be recorded.

Clinical parameters that will be recorded:

* EDSS score, a numeric value between 0 and 10
* Age, a numeric value > 18
* Disease duration, a numeric value (years)
* Sex, female or male

Standard Operating Procedures (SOPs)

Only the investigators will be responsible for data entry. As previously described, the analysis will be automated and checked for quality issues by researchers.

All data will be collected, encrypted, analyzed and stored on a dedicated sharepoint using the One Drive cloud service provided by the VUB, secured by password protection. All files from this server will be removed 5 years after the end of publication of the research results.

Sample size assessment

The investigators will use a one-tailed alpha of 0.05 (as the hypothesis is that worse visual scanning will relate to worse cognitive scores), a power of 0.8 (0.2 Type II error rate), and a correlation coefficient of 0.4 - corresponding to 16% of the variance of the SDMT being explained by eyesight - which leads to a sample size of 37. To be on the safe side and to account for possible data quality issues, the investigators will recruit N = 50 patients in this study.

Plan for missing data

In the exceptional case that some parameters are missing for some patients, those patients will be excluded from the specific analyses for which these datapoints are needed.

Statistical analyses plan

The correlation between eye movement parameters (VDI Pv/Am and VDI AUC, left and right), and cognitive test scores will be analyzed through Spearman correlation analysis.

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with clinically definite multiple sclerosis according to the 2017 McDonald criteria
* At least 18 years old
* Combined vision with optimal correction > 0,6 on Snellen Visual Acuity Test.
* Providing informed consent.

Exclusion criteria:

* Major medical or psychiatric pathology that potentially affects cognitive functioning.
* A score higher than 63 on the Fatigue Scale for Motor and Cognitive Functions is categorized as severe fatigue
* Start or switch in immunomodulatory treatment within three months before inclusion.
* Less than 3 months post exacerbation.
* Refusing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MS patients recruited from the neurology department of UZ Brussels and NMSC Melsbroek in Belgium
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between eye movement parameters and SDMT. | baseline
  Correlation between eye movement parameters (VDI AUC and VDI Pv/Am, left and right) and SDMT scores in patients with MS.

SECONDARY OUTCOMES:
Number of patients with eye movement abnormalities assessed by infrared oculography | Baseline
  The number of patients with VDI AUC>1.174 and/or VDI Pv/Am>1.180 assessed by infrared oculography during prosaccades at 15 degrees left or right.
Correlation between eye movement parameters and cognitive test scores. | Baseline
  The cognitive tests used to asses this correlation include the following: the PASAT (Paced Auditory Serial Addition Task), the CVLT-II (California Verbal Learning Test-II) and the BVMT-R (Brief Visuospatial Memory Test Revised).
  The correlation between eye movement parameters parameters (VDI Pv/Am and VDI AUC, left and right), and cognitive test scores will be analyzed through Spearman correlation analysis.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beier M, Gromisch ES, Hughes AJ, Alschuler KN, Madathil R, Chiaravalloti N, Foley FW. Proposed cut scores for tests of the Brief International Cognitive Assessment of Multiple Sclerosis (BICAMS). J Neurol Sci. 2017 Oct 15;381:110-116. doi: 10.1016/j.jns.2017.08.019. Epub 2017 Aug 16. PMID 28991659
- [Background] Meca-Lallana V, Gascon-Gimenez F, Ginestal-Lopez RC, Higueras Y, Tellez-Lara N, Carreres-Polo J, Eichau-Madueno S, Romero-Imbroda J, Vidal-Jordana A, Perez-Miralles F. Cognitive impairment in multiple sclerosis: diagnosis and monitoring. Neurol Sci. 2021 Dec;42(12):5183-5193. doi: 10.1007/s10072-021-05165-7. Epub 2021 Apr 1. PMID 33796947
- [Background] Van Schependom J, D'hooghe MB, Cleynhens K, D'hooge M, Haelewyck MC, De Keyser J, Nagels G. The Symbol Digit Modalities Test as sentinel test for cognitive impairment in multiple sclerosis. Eur J Neurol. 2014 Sep;21(9):1219-25, e71-2. doi: 10.1111/ene.12463. Epub 2014 May 22. PMID 24850580
- [Background] Nij Bijvank JA, Petzold A, Balk LJ, Tan HS, Uitdehaag BMJ, Theodorou M, van Rijn LJ. A standardized protocol for quantification of saccadic eye movements: DEMoNS. PLoS One. 2018 Jul 16;13(7):e0200695. doi: 10.1371/journal.pone.0200695. eCollection 2018. PMID 30011322
- [Background] Nij Bijvank JA, Hof SN, Prouskas SE, Schoonheim MM, Uitdehaag BMJ, van Rijn LJ, Petzold A. A novel eye-movement impairment in multiple sclerosis indicating widespread cortical damage. Brain. 2023 Jun 1;146(6):2476-2488. doi: 10.1093/brain/awac474. PMID 36535900
- [Background] Nij Bijvank JA, van Rijn LJ, Balk LJ, Tan HS, Uitdehaag BMJ, Petzold A. Diagnosing and quantifying a common deficit in multiple sclerosis: Internuclear ophthalmoplegia. Neurology. 2019 May 14;92(20):e2299-e2308. doi: 10.1212/WNL.0000000000007499. Epub 2019 Apr 19. PMID 31004067